CLINICAL TRIAL: NCT02444169
Title: Retrospective Evaluation of Safety of Combination Treatment With the Ulthera® System and Xeomin, Belotero Balance, and Radiesse
Brief Title: Retrospective Evaluation of Combination Treatment With the Ulthera System
Status: Completed | Type: Observational
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Other Study IDs: ULT-144
Record Dates: First submitted 2015-05-06; First posted 2015-05-14 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2015-08

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa | interventions — incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultherapy — Focused ultrasound energy delivered below the surface of the skin.
  Other Names: Ulthera System Treatment
Drug: Incobotulinumtoxin A — An injectable medicine used to temporarily improve the look of moderate to severe frown lines between the eyebrows (glabellar lines) in adults.
  Other Names: Xeomin
Device: Radiesse — An injectable dermal filler that temporarily adds volume to help smooth moderate to severe facial wrinkles and folds, such as nasolabial folds (the creases that extend from the corner of the nose to the corner of the mouth).
  Other Names: Volumizing filler
Device: Belotero Balance — An injectable dermal filler to temporarily smooth out and fill in moderate-to-severe nasolabial folds (the folds or wrinkles that go from the side of the nose to the corner of the mouth).
  Other Names: Dermal filler

SUMMARY:
A retrospective study to evaluate the Ulthera® System for its potential interaction with toxins and fillers. Up to 500 subjects will be enrolled.

DETAILED DESCRIPTION:
This is a retrospective, multi-site study involving chart reviews of subjects who have received an Ultherapy treatment along with Radiesse®, Xeomin®, and/or Belotero® Balance within six months apart in the face and/or neck areas. Enrolled subjects will have received an Ultherapy treatment along with botulinum toxin A and/or filler treatment(s) within the last two years and with filler and toxin treatment occurring within 6 months before or after Ultherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 25 to 70 years.
* Subject in good health
* Subject must have had an Ultherapy treatment and Merz branded neurotoxin/filler treatments within 6 months of one or more Ultherapy treatments.
* Subject must have had both Ultherapy and neurotoxin/filler within the last 2 years (since April 2013) and with toxin/filler treatment within 6 months proximity to the Ultherapy treatment date.
* Absence of physical or psychological conditions unacceptable to the investigator, especially those whom are contraindicated to receive treatments with Ultherapy, Belotero, Radiesse and/or Xeomin.
* Subjects who are identified with good photography, must have the ability to be contacted to provide authorization to disclose photographs for usage of previously taken photography, if photos are deemed worthy of publication.

Exclusion Criteria:

* Subjects who have had any and all Ultherapy treatment(s) before April 2013.
* Subjects who have not received Radiesse®, Xeomin®, and/or Belotero Balance® within 6 months of Ultherapy treatment date.
* Psychiatric drugs and/or diseases that in the investigators opinion would impair the subject from understanding the photo consent, if photos are chosen for publication.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults between 25 and 70 years of age who have received an Ultherapy treatment and toxin/filler within the last two years within six months apart and meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Within 6 months before or after Ultherapy
  An assessment of adverse events through chart review will evaluate the safety of combination treatments of Ultherapy with toxins/fillers.

CONTACTS AND LOCATIONS:
Overall Officials: Liss Misell, PhD, Study Director — Ulthera, Inc
Locations (5):
- United States (5):
  - Aesthetic Plastic Surgical Institute, Laguna Beach, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, San Diego, California
  - Skin Research Institute, Coral Gables, Florida
  - Maryland Laser Skin and Vein Institute, Hunt Valley, Maryland
  - Premier Clinical Research, Spokane, Washington